CLINICAL TRIAL: NCT02911558
Title: Implication of a Mobile Team of Palliative Care and Reality of the Palliative Approach in the Units
Acronym: EVE
Status: Terminated | Type: Observational
Why Stopped: Investigator's decision (departure from Institution)
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/68
Record Dates: First submitted 2016-09-13; First posted 2016-09-22 (Estimated); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Death; Palliative Care
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to estimate the impact of the implication of a Mobile Team of Palliative Care (EMSP) on the palliative strategy in the units with concerned patients. The Mobile Team of Palliative of Foch hospital Care was created in March, 2011.

ELIGIBILITY:
Inclusion Criteria:

* Patients died between July, 2013 and September, 2014 and for which at least one opinion of the EMSP was required

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients died between July, 2013 and September, 2014 and for which at least one opinion of the EMSP was required
Sampling Method: Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Time between specific treatments discontinuation and patient death | 6 months maximum

CONTACTS AND LOCATIONS:
Overall Officials: Edouard Ferrand, Principal Investigator — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France